CLINICAL TRIAL: NCT01641172
Title: Taste and Smell Changes in Testicular Cancer Patients Treated With Cisplatin Based Chemotherapy
Brief Title: Taste, Smell and Chemotherapy (TASTY)
Acronym: TASTY
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: University Medical Center Groningen (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: TASTY-01; NL38757.042.11 (Other: CCMO)
Record Dates: First submitted 2012-01-25; First posted 2012-07-16 (Estimated); Last update posted 2024-04-19 (Actual); Status verified 2024-04

CONDITIONS: Testicular Cancer
Keywords: taste; smell; cancer; nutrition
MeSH Terms: conditions — Testicular Neoplasms; Anosmia; Neoplasms | interventions — Absorptiometry, Photon; Hearing

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Patients (Active Comparator): Patients with disseminated testicular cancer
  Interventions: Procedure: Dexa scan; Procedure: audiogram; Procedure: measurement of heart rate variability and baroreflex sensitivity; Procedure: Glucose tolerance assessment; Dietary Supplement: oral nutrition supplements; Behavioral: Two day food records; Behavioral: Food Frequency Questionnaire
- Healthy volunteers (Placebo Comparator): Healthy men, age 18-50 years old
  Interventions: Procedure: Dexa scan; Procedure: audiogram; Procedure: measurement of heart rate variability and baroreflex sensitivity; Procedure: Glucose tolerance assessment; Dietary Supplement: oral nutrition supplements; Behavioral: Two day food records; Behavioral: Food Frequency Questionnaire

INTERVENTIONS:
Procedure: Dexa scan — the DEXA scan to measure bone and fat will be performed one time in the healthy controls and the patients participating in the cross sectional part of the study.
  The patients in the longitudinal part of the study will have a DEXA scan at baseline, 1 month after the end of chemotherapy and after 1 year.
  Other Names: Dual-energy X-ray absorptiometry
Procedure: audiogram — the audiogram will be performed one time in the healthy controls and the patients participating in the cross sectional part of the study.
  The patients in the longitudinal part of the study will have an audiogram at baseline, 1 month after the end of chemotherapy and after 1 year.
Procedure: measurement of heart rate variability and baroreflex sensitivity — the measurements (continuous assessment of heart rate and blood pressure using an non-invasive Finapress device) during 30 minutes will be performed one time in the healthy controls and the patients participating in the cross sectional part of the study.
  The patients in the longitudinal part of the study will have those measurements taken at baseline, 1 month after the end of chemotherapy and after 1 year.
  Other Names: HRV; BRS
Procedure: Glucose tolerance assessment — Glucose tolerance will be assessed by drinking glucose water and measuring glucose at baseline and 2 hours later. It will be performed one time in the healthy controls and the patients participating in the cross sectional part of the study.
  The patients in the longitudinal part of the study will have an assessment at baseline, 1 month after the end of chemotherapy and after 1 year.
Dietary Supplement: oral nutrition supplements — a set of 10 Oral Nutrition Supplements (ONS) will be offered combined with a questionnaire to measure appreciation and preference for these food products. All these tests and questionnaires will be performed longitudinally (before the first chemotherapy, on day 7 of the first course, before the second course, on day 7 of the second course, 1 month after start of the last course, 7 months after the start of chemotherapy, and 1 year after the start of chemotherapy) and cross-sectional (1, 3, 5 and 7 years after chemotherapy).
Behavioral: Two day food records — Two day food records will be used to investigate the actual dietary intake before the first and second course, during (on day 5 and 6) first and second course, 1 month after start of the last course, 7 months after the start of chemotherapy, and 1 year after the start of chemotherapy.
Behavioral: Food Frequency Questionnaire — A Food Frequency Questionnaire (FFQ) will be used to investigate the usual dietary intake before the start of the first course, before and after the second course, 1 month after start of the last course, seven months after the start of chemotherapy, and 1 year after the start of chemotherapy (longitudinal), and 1, 3, 5 and 7 years after chemotherapy (cross-sectional).
  Other Names: FFQ

SUMMARY:
Taste and smell abnormalities are common in cancer patients undergoing chemotherapy, with a prevalence ranging from 46% to 77% for taste changes, and 35% to 75% for smell changes. These chemosensory changes are distressing for patients and can lead to changes in appetite, food choice, and nutrient intake. These changes can result in malnutrition and weight loss. Possibly, also unhealthy eating patterns can be developed due to these taste and smell changes, given the high prevalence of obesity among survivors of certain cancer types. The primary objective is to investigate the nature, prevalence, and duration of taste and smell changes in patients with disseminated testicular cancer treated with cisplatin based chemotherapy.

DETAILED DESCRIPTION:
Rationale: Taste and smell abnormalities are common in cancer patients undergoing chemotherapy, with a prevalence ranging from 46% to 77% for taste changes, and 35% to 75% for smell changes. These chemosensory changes are distressing for patients and can lead to changes in appetite, food choice, and nutrient intake. These changes can result in malnutrition and weight loss. Possibly, also unhealthy eating patterns can be developed due to these taste and smell changes, given the high prevalence of obesity among survivors of certain cancer types. Objective: The primary objective is to investigate the nature, prevalence, and duration of taste and smell changes in patients with disseminated testicular cancer treated with cisplatin based chemotherapy. Secondary objectives are to explore the short- and long-term consequences of these chemosensory changes for (medical) food preference, dietary intake and quality of life, and to investigate the appreciation of medical food products in these testicular cancer patients. Furthermore, it will be assessed whether changes in taste and smell are related to the metabolic syndrome, and whether chemotherapy induced neurotoxicity is related to changes in taste and smell. Study design: The present study will have a longitudinal (with measurements before the first chemotherapy, on day 7 of the first course, before the second course, on day 7 of the second course, 1 month after start of the last course, 7 months after the start of chemotherapy, and 1 year after the start of chemotherapy) and a cross-sectional (with measurements 1, 3, 5 and 7 years after chemotherapy) design. Patients can start participation in this study before the start of their chemotherapy, which will result in longitudinal data of these patients or they can start participation years after treatment, resulting in cross-sectional data.

Study population: Patients with disseminated testicular cancer treated with cisplatin based chemotherapy. This group is selected, because of the young age at diagnosis, the emetogenic chemotherapy treatment, the high survival rate, the increase in body mass index (BMI) and risk of cardiovascular disease in the long-term.

Intervention: Gustatory function will be tested using filter-paper taste strips to measure recognition thresholds for sweet, salty, sour and bitter taste. Olfactory function will be tested using Sniffin' Sticks to measure odor threshold, discrimination and recognition.

Besides, patients have to fill out questionnaires to assess taste and smell subjectively and to assess QoL. Food preference will be investigated by showing standardized photographs of sweet and savory food products, varying in fat and protein content. In addition, a set of 10 Oral Nutrition Supplements (ONS) will be offered combined with a questionnaire to measure appreciation and preference for these food products. All these tests and questionnaires will be performed longitudinally (before the first chemotherapy, on day 7 of the first course, before the second course, on day 7 of the second course, 1 month after start of the last course, 7 months after the start of chemotherapy, and 1 year after the start of chemotherapy) and cross-sectional (1, 3, 5 and 7 years after chemotherapy). Two day food records will be used to investigate the actual dietary intake before the first and second course, during (on day 5 and 6) first and second course, 1 month after start of the last course, 7 months after the start of chemotherapy, and 1 year after the start of chemotherapy. A Food Frequency Questionnaire (FFQ) will be used to investigate the usual dietary intake before the start of the first course, before and after the second course, 1 month after start of the last course, seven months after the start of chemotherapy, and 1 year after the start of chemotherapy (longitudinal), and 1, 3, 5 and 7 years after chemotherapy (cross-sectional).

A Dual Energy X-ray Absortiometrys (DEXA) scan will be used to get insight in possible changes in bone and fat mass during and after chemotherapy. To detect a possible cause of taste and smell changes, audiogram will be performed (to measure cisplatin induced neurotoxicity), and the baroreflex sensitivity (BRS) (to measure the quality of shortterm blood pressure maintenance), the blood glucose tolerance, insulin resistance, and DNA for SNP analysis will be collected. The DEXA scan, audiogram, BRS test, and blood glucose tolerance test will be performed before the first course of chemotherapy, one month after start of the last course, 1 year after the start of chemotherapy (longitudinal part), and 1, 3, 5 and 7 years after chemotherapy (cross-sectional part). A blood sample for DNA analysis will be taken at the start of the chemotherapy (longitudinal part), and 1, 3, 5 and 7 years after chemotherapy (cross-sectional part).

ELIGIBILITY:
Inclusion Criteria:

* Patients with disseminated testicular cancer undergoing first line cisplatin based chemotherapy (BEP or EP).
* Age 18-50 years at start of treatment.
* Signed informed consent.
* Ability to comprehend Dutch (both reading and writing).
* Complete remission after cisplatin based chemotherapy (BEP or EP) with or without adjunctive surgery and in active follow-up (only for crosssectional part of the study).

Exclusion Criteria:

* Mental disability
* Patients with co-morbidities that affect gustatory or olfactory function, such as rhinosinusitis, liver or renal problems, hyperactivity or hypoactivity of the thyroid gland, diabetes, or neurologic disorders (only for crosssectional part of the study).

Ages: 18 Years to 50 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 140 (Actual)
Dates: Start 2012-06; Primary Completion 2016-01 (Actual); Study Completion 2016-01 (Actual)

PRIMARY OUTCOMES:
investigate the nature, prevalence, and duration of taste and smell changes | baseline, day 7 of first course, before 2nd course, day 7 2nd course, 1 month after start of last course, 7 months after start of chemotherapy, 1 year after start study; 1, 3, 5 and 7 years after chemotherapy.
  To investigate the nature, prevalence, and duration of taste and smell changes in patients with disseminated testicular cancer treated with cisplatin based chemotherapy (BEP (Bleomycin, Etoposide, cisPlatin) or EP (Etoposide, cisPlatin)).
  Tests used are: Gustatory function will be tested using filter-paper taste strips to measure recognition thresholds for sweet, salty, sour and bitter taste. Olfactory function will be tested using Sniffin' Sticks to measure odor threshold, discrimination and recognition.

SECONDARY OUTCOMES:
explore the short- and long-term consequences of taste and smell changes | baseline, day 7 of first course, before 2nd course, day 7 2nd course, 1 month after start of last course, 7 months after start of chemotherapy, 1 year after start study; 1, 3, 5 and 7 years after chemotherapy.
  To explore the short- and long-term consequences of taste and smell changes in relation to food preference, dietary intake, and quality of life. Tests used: QoL questionnaires (EORTC QLQ-C30). Two day food records will be used to investigate the actual dietary intake before the first and second course, during (on day 5 and 6) first and second course, 1 month after start of the last course, 7 months after the start of chemotherapy, and 1 year after the start of chemotherapy. A Food Frequency Questionnaire (FFQ) will be used to investigate the usual dietary intake.
investigate the appreciation of medical food products | baseline, day 7 of first course, before 2nd course, day 7 2nd course, 1 month after start of last course, 7 months after start of chemotherapy, 1 year after start study; 1, 3, 5 and 7 years after chemotherapy.
  To investigate the appreciation of medical food products in patients with disseminated testicular cancer treated with cisplatin based chemotherapy.
  A set of 10 Oral Nutrition Supplements (ONS) will be offered combined with a questionnaire to measure appreciation and preference for these food products.
  Food preference will be investigated by showing standardized photographs of sweet and savory food products, varying in fat and protein content.
Are changes related to metabolic syndrome? | baseline, 1 month after start of last course, 1 year after start study; 1, 3, 5 and 7 years after chemotherapy.
  To assess whether changes in taste and smell are related to the metabolic syndrome.
  Tests used: glucose tolerance test and DEXA scan.
Is chemotherapy induced neurotoxicity related to changes? | baseline, 1 month after start of last course, 1 year after start study; 1, 3, 5 and 7 years after chemotherapy.
  To assess whether chemotherapy induced neurotoxicity is related to changes in taste and smell.
  TEsts used: audiogram, assessment of heart rate variability and baroreflex sensitivity.

CONTACTS AND LOCATIONS:
Overall Officials: A KL Reyners, MD, PhD, Principal Investigator — University Medical Center Groningen
Locations (1):
- University Medical Center Groningen, Groningen, Netherlands